CLINICAL TRIAL: NCT06135116
Title: CD4+CD25+High FOXp3+ Regulatory T Cell With Related Interleukins and Vitamin D-binding Protein in Periodontal Disease Progression : Synergy or Cocaphony
Brief Title: Regulatory T Cell With Related Interleukins in Periodontal Disease Progression
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, lecturer ,Oral medicine and periodontology, Al-Azhar University
Other Study IDs: Treg in periodontitis
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis; Gingivitis
Keywords: inflammation; Periodontitis; Cytokines; Vitamin D-Binding Protein; Interleukin-33; nterleukin-21
MeSH Terms: conditions — Periodontitis; Gingivitis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- periodontally healthy: twenty persons without any signs of periodontal disease. This was determined by the absence of attachment loss and bleeding upon probing either ˂ 10% or probing depth ˂3 mm.
  Interventions: Diagnostic Test: Flow Cytometric Detection of Regulatory T Cells and Cytokines analysis by ELISA
- chronic gingivitis: twenty persons exhibiting generalized chronic gingivitis exhibiting signs of erythema, bleeding on probing up to 20%, edema, probing pocket depth less than 3 mm and no periodontal attachment loss.
  Interventions: Diagnostic Test: Flow Cytometric Detection of Regulatory T Cells and Cytokines analysis by ELISA
- chronic periodontitis: twenty patients having severe generalized form of chronic periodontitis exhibiting PPD ≥ 6 mm, CAL ≥ 5mm and bone loss affecting at least six teeth as observed in dental periapical radiograph
  Interventions: Diagnostic Test: Flow Cytometric Detection of Regulatory T Cells and Cytokines analysis by ELISA

INTERVENTIONS:
Diagnostic Test: Flow Cytometric Detection of Regulatory T Cells and Cytokines analysis by ELISA — Gingival crevicular fluid samples collection After removing supragingival plaque, sampling sites were isolated by cotton rolls and dried using air syringe, GCF samples were collected by inserting standardized paper point in the sulcus/ pocket at the proximal-facial line angle of six preselected sites in each patient teeth . Fluid was sucked by paper points for 30 seconds. The samples were immediately placed inside graduated eppendorf vials containing 250µl phosphate-buffered saline (PBS), and transported to the laboratory for subsequent assays .
  Blood Samples Collection From control and patient groups and under standard aseptic conditions, the peripheral blood was collected in Ethelene Diamine Tetra Acetic Acid (EDTA) coated vacutainer tubes (K2 EDTA) 5.4mg (BD vacutainer) and transferred immediately to flow cytometric analysis lab.

SUMMARY:
T Regulatory cells which suppressor subset of T cells and related cytokines remain in blood and infiltrates into the tissue under need. The role of Treg and related cytokines in succession of periodontal inflammation is recently a subject of research interest. Chronic gingivitis and periodontitis being chronic inflammatory diseases can upregulate various cytokines in the systemic circulation and gingival crevicular fluid. This study aimed to compare levels of Tregs with Interleukin-21, 22, 33, 35 and vitamin D-binding protein in blood and GCF of periodontally healthy persons, chronic gingivitis patients, and severe chronic periodontitis patients.

DETAILED DESCRIPTION:
T regs infiltration might reveal a trial to control tissue damage, however it also might be suggestive of a destructive effect of Tregs in periodontitis . Tregs can actually play a damaging role as this cells can annoyingly weaken the immune reaction towards infectious agents that could be possibly harmful in a periodontal environment . Immunopathology of Treg cell mediated via its pro-inflammatory cytokines during inflammatory conditions. IL-33 "recent member of pro-inflammatory IL-1 category" was recognized as placard in the stability of Foxp3+ Treg cell at mucosal sites. IL-33 has either pro- or anti-inflammatory property according to the disease and the model. It was speculated that IL-33 could improve the propagation from suppressive to dysregulated Treg cells in a dose-dependent manner . Interleukin (IL)-21 which member of the type I (ℽ chain) cytokine family has the ability to minimize FoxP3 expression and restraining Treg suppressor function and homeostasis . The purpose from this study was to assess the role of circulating and localized Treg with their related cytokines in patients with inflammation of periodontal tissues and to correlate their levels with disease progression.

ELIGIBILITY:
Inclusion Criteria:

* periodontally healthy persons without any signs of periodontal disease. This was determined by the absence of attachment loss and bleeding upon probing either ˂ 10% or probing depth ˂3 mm.
* persons exhibiting generalized chronic gingivitis exhibiting signs of erythema, bleeding on probing up to 20%, edema, probing pocket depth less than 3 mm and no periodontal attachment loss.
* persons having severe generalized form of chronic periodontitis exhibiting PPD ≥ 6 mm, CAL ≥ 5mm and bone loss affecting at least six teeth as observed in dental periapical radiograph.

Exclusion Criteria:

* Patients with systemic diseases according to Modified Cornell Medical Index criteria
* Patients receiving either antibiotics or non-steroidal anti- inflammatory at least 3 months prior to samples collection.
* Patients subjected to previous periodontal therapy 6 months before sampling.
* Patients with systemic or local inflammatory conditions other than periodontal disease.
* The smokers.
* Neither lactating nor pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty persons will be selected from the attendance of the out-patient clinic, Oral Medicine and Periodontology Department, Faculty of Dentistry, Al-Azhar University, Assiut. They divided according to the periodontal health status into three groups.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Treg cells frequency | baseline(through clinical diagnosis completion)
  evaluation of frequency of systemic and GCF levels of T regs in patients (periodontitis and gingivitis) and healthy group.Regulatory T cells were quantitively estimated using fluoroisothiocyanate (FITC)-conjugated Foxp3 (e Bioscience, USA), phycoerythrin (PE) conjugated CD25 (IQ Product, The Netherland) and peridinium-chlorophyll-protein (Per-CP)-conjugated CD4 (Becton Dickinson, Bioscience, USA).
Cytokines levels (IL-22, IL-21, IL-35, IL-33) and vitamin D binding protien | baseline(through clinical diagnosis completion)
  comparative evaluation of systemic and GCF levels of cytokines in different periodontal conditions; healthy, gingivitis and periodontitis.they were measured by a commercially available enzyme-linked immunosorbent assay kits as following; ELISA kit (Legend Max, BioLegend, San Diego, CA, USA) with undetectable level below 20 pg/ml for IL-21, ELISA kit (RayBiotech. Norcross, Georgia, USA) with undetectable level below 8 pg/ml for IL-22, ELISA kit (GenWay Biotech Inc. San Diego, CA, USA) with undetectable level below 0.7ng/ml for IL-33, ELISA kit (Glory Science CO., Ltd, Del Rio, TX, USA) for IL-35 and finally ELISA kit (BioSource Systems, Invitrogen, Grand Island, NY, USA) for DBP.

SECONDARY OUTCOMES:
dental Plaque score | baseline(through clinical diagnosis completion)
  measured by O'Leary Plaque score as following; bacterial deposits where be stained with a disclosing solution to facilitate their detection. Calculation = the number of plaque containing surfaces / the total number of available surfaces. In the rating system, 0% indicates absence of plaque, with 15 %, 20 %, and > 40% indicating an increased percentage of plaque accumulation.
Bleeding on probing (BoP) | Baseline(through clinical diagnosis completion)
  By a force of 0.25 N. by a manual pressure of sensitive probe, recorded on distal, facial, mesial, gingival surfaces. Bleeding on probing (BoP) Calculated as following; Number of bleeding surfaces / total number of tooth surface) multiplying in one hundred and expressed in percentage (%). In the rating system, 0 indicates absence of bleeding on probing (healthy), with 15%, 20% (gingivitis) and >20% indicating an increased percentage of inflammation/infection (periodontitis).
Probing pocket depth | Baseline(through clinical diagnosis completion)
  it was measured from the gingival margin to the base of the pocket by William's graduated periodontal probe
Attachment level | Baseline(through clinical diagnosis completion)
  it was measured by subtracting the distance from the cemento-enamel junction to the free gingival margin from the distance from the free gingival margin to the base of the pocket both were properly measured using William's graduated probe and the difference between the two measurements yields the attachment level

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral medicine, Periodontology, Oral diagnosis and dental radiology Faculty of dental medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Meng H, Sun X, Xu L, Zhang L, Shi D, Feng X, Lu R, Chen Z. Elevation of vitamin D-binding protein levels in the plasma of patients with generalized aggressive periodontitis. J Periodontal Res. 2013 Feb;48(1):74-9. doi: 10.1111/j.1600-0765.2012.01505.x. Epub 2012 Jul 18. PMID 22803589
- [Background] Nakajima T, Ueki-Maruyama K, Oda T, Ohsawa Y, Ito H, Seymour GJ, Yamazaki K. Regulatory T-cells infiltrate periodontal disease tissues. J Dent Res. 2005 Jul;84(7):639-43. doi: 10.1177/154405910508400711. PMID 15972593
- [Background] Hasan A, Palmer RM. A clinical guide to periodontology: pathology of periodontal disease. Br Dent J. 2014 Apr;216(8):457-61. doi: 10.1038/sj.bdj.2014.299. PMID 24762896